CLINICAL TRIAL: NCT05356520
Title: A Multicenter Randomized Controlled Study of Siewert II Esophagogastric Junction Adenocarcinoma With Endoscopic Ivor-Lewis Approach Versus Laparoscopic Transabdominal Extended Gastrectomy
Brief Title: Comparison of Different Operations for Siewert Type II Adenocarcinoma of Esophagogastric Junction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Tang-Du Hospital (Other); Henan Provincial People's Hospital (Other); General Hospital of Ningxia Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, xiaohua li, Associate chief physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJ MZC 2022 04
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Siewert Type II Adenocarcinoma of Esophagogastric Junction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): Endoscopic ivor-Lewis operation was performed for siwert type II adenoma at the esophagogastric junction
  Interventions: Procedure: Endoscopy Ivor-lewis
- The control group (Active Comparator): Laparoscopic transabdominal enlarged gastrectomy for siwert TYPE II adenoma at the esophagogastric junction was performed
  Interventions: Procedure: Laparoscopic transabdominal enlarged gastrectomy

INTERVENTIONS:
Procedure: Endoscopy Ivor-lewis — Endoscopy Ivor-lewis
  Arms: The experimental group
Procedure: Laparoscopic transabdominal enlarged gastrectomy — Laparoscopic transabdominal enlarged gastrectomy
  Arms: The control group

SUMMARY:
The incidence of esophagogastric junction has been increasing in recent years, and surgery is an important method for the treatment of adenoma at the esophagogastric junction. Currently, there is a great controversy about the surgical method of Siewert II, mainly choosing the right chest or the left chest for thoracic surgery. Therefore, it is of great significance to further study the surgical methods of Siewert II esophagogastric junction adenoma. Objective: To compare the safety, feasibility, and clinical efficacy of endoscopic Ivor-Lewis versus laparoscopic extended abdominal gastrectomy for Siewert type Ⅱadenocarcinoma at the resectable esophagogastric junction.

DETAILED DESCRIPTION:
At present, the main surgical approaches for the treatment of esophagogastric junction adenocarcinoma include single left thoracic incision, 2 right epigastric incisions, 2 left epigastric incisions, 3 cervicothoracoabdominal incisions, and left thoracoabdominal combined incision and esophageal rift through the diaphragm. Siewert type I ESOPHAgogastric junction carcinoma recommends a right thoracic approach, including Ivor-LEIws and McKeown, according to the Chinese Expert consensus for surgical treatment of ESOPHAgogastric junction adenocarcinoma published in 2018. Siwert TYPE III adenoma at esophagogastric junction, esophageal hiatus through diaphragmatic approach is recommended. The surgical approach for siwert type II adenoma at the esophagogastric junction is controversial [7,8]. Due to the particularity of siWERT type II lymph node diffusion, it can spread to both posterior mediastinal lymph nodes and abdominal lymph nodes, and a simple esophageal hiatus through the diaphragm may not be enough to clear lymph nodes. Does a combined thoracoabdominal approach improve patient outcomes? In the 1990s and early 2000s, the Japanese Clinical Oncology Organization (JCOG) compared the efficacy of different surgical approaches for esophagogastric junction adenocarcinoma. The trial randomized patients to transesophageal hiatus or left thoracoabdominal combined approach. Results The incidence of postoperative pneumonia was significantly higher in the left thoracoabdominal approach group than in the transesophageal hiatus group (13%vs. 4%, P=0.048), there was no significant difference in the survival rate of Siewert II type ESOPHAgogastric junction tumor between the two groups (P=0.496). To provide the best, targeted treatment for patients with esophagogastric junction adenocarcinoma, radical resection of the tumor should be combined with resection of adjacent lymph nodes. Previous studies have shown that the effect of surgery on the right chest is better than that on the left. Therefore, we asked whether the endoscopic Ivor-Lewis approach was better than the laparoscopic transabdominal enlarged gastrectomy. The right thoracic approach is the recommended approach for siwert type I adenoma at the esophagogastric junction. It has obvious advantages in postoperative esophageal and cardiopulmonary function protection. Currently, there are no clinical trials of endoscopic Ivor-Lewis and laparoscopic extended abdominal gastrectomy for the treatment of siwert type II adenoma at the esophagogastric junction. Endoscopic IVOR-Lewis and laparoscopic transesophageal hiatus test provide new clinical data for the treatment of siwert TYPE II adenoma at the esophagogastric junction, and help standardize the treatment of siwert type II adenoma at the esophagogastric junction. Therefore, based on our experience and foundation of gastrointestinal surgery in the treatment of esophagogastric junction tumors, through practical observation and research on clinical experimental treatment plans, and integration of domestic superior resources, the establishment and improvement of treatment standards for esophagogastric junction adenoma will be further promoted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed EGJ type II adenocarcinoma

  ··The tumor can be removed by laparoscopy through the gastrodiaphragmatic esophageal hiatus or by endoscopic Ivor Lewis operation
* Pretreatment stage CT1-4A, N0-3, M0
* For cT4a stage patients, their resectable properties must be clearly verified before randomization
* For locally advanced tumors (CT3-T4 or N+), all 4 cycles of chemotherapy (FLOT) were completed before surgery.
* 18 to 75 years old
* ECOG score 0-2
* ASA <4
* Good bone marrow function (leukocyte > x 10 ^ 9 / l; Hemoglobin> 9 g/dl. ·Platelet>100×10^9/ L), renal function (glomerular filtration rate & GT; 60ml/min) and liver function (total bilirubin < 1.5 times normal (ULN), aspartate aminotransferase (AST< 2.5x ULN, Alanine aminotransferase (ALT)<3 x ULN)
* Patients and their family members voluntarily sign written informed consent

Exclusion Criteria:

* Histologically confirmed EGJ type I and III adenocarcinoma
* Tumor spread over 5 cm proximal to EGJ
* Clinically significant (active) heart disease (i.e. symptomatic coronary artery disease or myocardial infarction within the last 12 months) resulting in left ventricular ejection fraction<50%(determined by echocardiography)
* Clinically significant lung diseases (forced expiratory volume in 1 second (FEV1)<1.5 l/s)
* Pregnant women and nursing mothers
* Stump gastric cancer
* Borrmann Type 4 (Leather stomach)
* Simultaneous or heterochronous malignant tumors of other organs except carcinoma in situ of the cervix and adenoma and focal colorectal carcinoma
* Right thoracotomy or history of right pleural adhesion
* Cirrhosis, or indocyanine green test ≥15% of chronic liver disease
* No seizure control, central nervous system diseases or mental disorders
* History of upper abdominal surgery (except laparoscopic cholecystectomy)
* The patient has coagulation dysfunction and cannot be corrected
* Patients with heart, lung, liver, brain, kidney and other important organ failure
* Patients with metabolic diseases such as diabetes
* Immunosuppressive therapy, such as organ transplantation, SLE, etc
* Seriously out of control recurrent infections or other seriously out of control concomitant diseases
* Other diseases requiring simultaneous surgery
* Diseases requiring emergency surgery due to tumor emergencies (e.g. hemorrhage, perforation, obstruction)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | three years
  The time from the date of surgery to the patient's death from any cause

SECONDARY OUTCOMES:
Overall survival | five years
  The time from the date of surgery to the patient's death from any cause
Incidence of postoperative complications | a month
  Postoperative complications include anastomotic fistula (clinically or radiologically diagnosed); Respiratory complications (defined as clinical manifestations of pneumonia or bronchopneumonia, confirmed by computed tomography); Cardiovascular complications (defined as persistent arrhythmias requiring treatment); Chylothorax (defined as white fluid in thoracic drainage after enteral nutrition); Wound infection; And other complications (delayed empty. pleural effusion, recurrent nerve injury)
Postoperative mortality | a month
  Postoperative mortality is defined as the proportion of deaths from any cause
Tumor recurrence | three years
  Tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: xiaohua li, MD,PH.D, Study Chair — Xijing Hospital; xianli he, MD,PH.D, Principal Investigator — Tang-Du Hospital; peichun sun, MD,PH.D, Principal Investigator — Henan Provincial People's Hospital; lei wang, MD,PH.D, Principal Investigator — General Hospital of Ningxia Medical University; xuejun sun, MD,PH.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; he huang, MD,PH.D, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University
Locations (1):
- Li, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yue C, Mo Z, Wu X, Wang Y, Yang Q, Wang W, Zhou H, Gao R, Ji P, Dong D, Zhang Y, Ji G, Li X. Comparison of thoracoabdominal versus abdominal-transhiatal surgical approaches in Siewert type II adenocarcinoma at the esophagogastric junction: Protocol for a prospective multicenter randomized controlled trial. Front Oncol. 2023 Mar 30;13:1091615. doi: 10.3389/fonc.2023.1091615. eCollection 2023. PMID 37064105